CLINICAL TRIAL: NCT06398145
Title: The Use of D-chiro-inositol in the Treatment of AUB
Brief Title: D-chiro-inositol and AUB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Sandro Gerli, Professor, University Of Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INOSENDO
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Lactalbumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will undergo 3 months treatment with 1200 mg D-chiro-inositol and 120 mg lactalbumin, than 3 months treatment with 600 mg D-chiro-inositol and 60 mg lactalbumin
  Interventions: Dietary Supplement: D-chiro-inositol and lactalbumin (high dose); Dietary Supplement: D-chiro-inositol and lactalbumin (low dose)

INTERVENTIONS:
Dietary Supplement: D-chiro-inositol and lactalbumin (high dose) — From 0 to 3 months: 1200mg D-chiro-inositol and 120mg lactalbumin per day
Dietary Supplement: D-chiro-inositol and lactalbumin (low dose) — From 3 to 6 months: 600mg D-chiro-inositol and 60mg lactalbumin per day

SUMMARY:
Patients with AUB will undergo 6-month treatment with D-chiro-inositol and will fill in questionnaires on AUB, with the evaluation of hormonal serum levels.

ELIGIBILITY:
Inclusion Criteria:

* AUB

Exclusion Criteria:

* Menopause
* Cancer diagnosis
* Atypical endometrial hyperplasia
* Uterine fibroids
* Heavy symptoms requiring pharmacological intervention
* Progestogens treatment in the six months before the study
* Inositol treatment in the six months before the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
AUB | 0, 3 and 6 months
  The "Menstrual Bleeding Questionnaire", a standardized and validated questionnaire, will be administered to patients to evaluate te extent of AUB and the impact on their quality of life.

SECONDARY OUTCOMES:
Serum level of Estradiol | 0, 3 and 6 months
  Serum levels of estradiol will be evaluated after intravenous blood sampling
Serum level of Estrone | 0, 3 and 6 months
  Serum levels of estrone will be evaluated after intravenous blood sampling
Serum level of Testosterone | 0, 3 and 6 months
  Serum levels of testosterone will be evaluated after intravenous blood sampling
Serum level of Androstenedione | 0, 3 and 6 months
  Serum levels of androstenedione will be evaluated after intravenous blood sampling
Serum level of Total cholesterol | 0, 3 and 6 months
  Serum levels of total cholesterol will be evaluated after intravenous blood sampling
Serum level of High-Density Lipoprotein | 0, 3 and 6 months
  Serum levels of HDL will be evaluated after intravenous blood sampling
Serum level of Low-Density Lipoprotein | 0, 3 and 6 months
  Serum levels of LDL will be evaluated after intravenous blood sampling
Serum level of Triglyceride | 0, 3 and 6 months
  Serum levels of triglyceride will be evaluated after intravenous blood sampling